CLINICAL TRIAL: NCT02206685
Title: A Randomized Blinded Prospective Trial Comparing Single Intraoperative Dose of Methadone Versus Placebo in Pediatric Patients Undergoing Spine Surgery.
Brief Title: A Trial Comparing Single Intra-op Dose of Methadone Versus Placebo in Patients Undergoing Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kim Nguyen, Pediatric Anesthesiologist, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H32894
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Thoracolumbar Scoliosis
MeSH Terms: interventions — Methadone; Saline Solution; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Active Comparator): The treatment group will receive 0.2 mg/kg methadone diluted to a 20 ml infusion over 10 minutes.
  Interventions: Drug: Methadone
- Control Group (Placebo Comparator): The control group will receive a 20 ml normal saline placebo infusion over 10 minutes
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Methadone — The treatment group will receive 0.2 mg/kg methadone diluted to a 20 ml infusion over 10 minutes
  Other Names: Treatment group
  Arms: Treatment group
Drug: Normal Saline — the control group will receive a 20 ml normal saline placebo infusion over 10 minutes
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
Scoliosis is a disease that involves lateral and/or rotational deformity of the spine and can affect up to 4% of the population. Typically, surgery is considered when Cobb's angle, which is a measurement used for evaluation of curves in scoliosis on an anterior-posterior radiographic projection of the spine, is greater than 50 degrees in the thoracic region (40 degrees in the lumbar region) or when the curvature causes significant pain, or respiratory and cardiovascular restriction. Patient undergoing this surgical correction experience severe pain in the postoperative period and the management includes the use of opioid-based patient-controlled analgesia (PCA).

DETAILED DESCRIPTION:
Scoliosis is a disease that involves lateral and/or rotational deformity of the spine and can affect up to 4% of the population. Typically, surgery is considered when Cobb's angle, which is a measurement used for evaluation of curves in scoliosis on an anterior-posterior radiographic projection of the spine, is greater than 50 degrees in the thoracic region (40 degrees in the lumbar region) or when the curvature causes significant pain, or respiratory and cardiovascular restriction. Patient undergoing this surgical correction experience severe pain in the postoperative period and the management includes the use of opioid-based patient-controlled analgesia (PCA).

Methadone is an opioid with one of the longest elimination half-life and has been used as an effective analgesic for acute, chronic, neuropathic, and cancer pain in adults, children, and even neonates1-5. Its long duration of action and antagonism to the N-methyl-d-aspartate receptor may decrease the need for PCA use in the postoperative period. Gourlay2 demonstrated the effectiveness and utility of perioperative methadone including the advantages of longer analgesia with no serious side effects of respiratory depression. A recent study by Gottschalk2 in adult patients demonstrated a 50% reduction of postoperative opioids at 48 hours and lower pain scores after a single bolus of methadone before surgical incision. However, a major weakness of the study is that patients did not receive equipotent intraoperative opioids. In addition, the adolescent patient population will undergo a much larger surgical incision with potential for greater postoperative pain. Despite this potential benefit, methadone is seldom used in the perioperative setting. A more recent pharmacokinetic study of methadone in adolescents undergoing spine surgery failed to show a reduction in opioid consumption as it was powered to determine pharmacokinetics and not a secondary endpoint of postoperative opioid consumption. An appropriately powered study is still required to determine the efficacy of methadone in reducing postoperative pain after spine surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 10 - 17 years
2. Patients undergoing multilevel thoraco-lumbar spine surgery with instrumentation and fusion

Exclusion Criteria:

1. Preoperative methadone therapy
2. Inability to use the PCA
3. Allergy to methadone or morphine
4. Morbid obesity with a body mass index >36.0 kg/m2
5. Patients with chronic renal failure defined by serum creatinine >2.0 mg/dL
6. Liver failure defined as a history of cirrhosis or fulminant hepatic failure
7. Preoperative congenital heart disease or arrhythmias
8. Patient refusal to participate in study
9. Pregnancy (It is standard of care for all post menarche female patients to undergo a urine pregnancy test prior to surgery).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Nguyen, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Methods of statistical analysis may be shared at study completion.

REFERENCES:
- [Background] Nicholson AB. Methadone for cancer pain. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003971. doi: 10.1002/14651858.CD003971.pub3. PMID 17943808
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Sharma A, Tallchief D, Blood J, Kim T, London A, Kharasch ED. Perioperative pharmacokinetics of methadone in adolescents. Anesthesiology. 2011 Dec;115(6):1153-61. doi: 10.1097/ALN.0b013e318238fec5. PMID 22037641
- [Background] Berde CB, Beyer JE, Bournaki MC, Levin CR, Sethna NF. Comparison of morphine and methadone for prevention of postoperative pain in 3- to 7-year-old children. J Pediatr. 1991 Jul;119(1 Pt 1):136-41. doi: 10.1016/s0022-3476(05)81054-6. PMID 2066846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 37 | 37
Completed | 32 | 30
Not Completed | 5 | 7
Not completed — Surgery cancelled/changed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.09 (1.69) | 14.33 (1.69) | 14.21 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62
Weight [Mean (Standard Deviation); unit: kg] | 58.26 (12.72) | 53.95 (13.20) | 56.18 (12.92)
Height [Mean (Standard Deviation); unit: cm] | 160.64 (9.98) | 162.48 (8.07) | 161.53 (9.01)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.45 (3.78) | 20.29 (3.89) | 21.41 (3.92)
ASA Status [Count of Participants; unit: Participants] — The ASA (American Society of Anesthesiologists) physical status classification system is a system for assessing the fitness of patients before surgery.
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease
  Participants
    I | 7 | 3 | 10
    II | 22 | 27 | 49
    III | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Opioid Usage
Description: Subjects were given access to Patient-Controlled Intravenous Opioid Administration (PCA) to manage their post-operative pain. The doses of morphine were calculated at at PACU, 24 hours, 48 hours and 72 hours respectively.
Time Frame: Admission to PACU to 72 hours post-operative
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 32 | 30
mg/kg
  PACU | 0.41 [0.25 to 0.65] | 0.47 [0.33 to 0.62]
  24 Hours | 0.58 [0.34 to 0.82] | 0.55 [0.37 to 0.66]
  48 Hours | 0.58 [0.31 to 0.79] | 0.55 [0.24 to 0.65]
  72 Hours | 0.10 [0 to 0.23] | 0.04 [0 to 0.14]

2. Secondary Outcome: Pain Scores
Description: The FLACC scale or Face, Legs, Activity, Cry, Consolability scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. The data reported here represents the mean difference in FLACC score by treatment group at PACU, 24 hours, 48 hours and 72 hours, respectively.
Time Frame: Admission to PACU to 72 hours post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 32 | 30
units on a scale
  PACU | 0.53 (0.76) | 0.65 (0.70)
  24 Hours | 0.14 (0.4) | 0.42 (0.66)
  48 Hours | 0.24 (0.45) | 0.36 (0.62)
  72 Hours | 0.16 (0.18) | 0.29 (0.64)

ADVERSE EVENTS:
Time Frame: At any time during hospitalization (Days 0 to 5)
Description: Side effects of Methadone versus Placebo group were assessed during the duration of the subject's hospitalization. Incidents were counted once per subject.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 15/32 | 14/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=32) | Control Group (N=30)
Nausea and Vomiting (Gastrointestinal disorders) | 15 | 14
Constipation (Gastrointestinal disorders) | 0 | 3
Hypoxemia (oxygen required) (Respiratory, thoracic and mediastinal disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT02206685/Prot_SAP_000.pdf